CLINICAL TRIAL: NCT02250144
Title: Foot Orthoses in Patellofemoral Pain Syndrome: a Prospective Randomized Study of Morpho-specific Versus Placebo Orthoses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5832
Record Dates: First submitted 2014-09-16; First posted 2014-09-26 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome; Feet orthoses; KOOS
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morpho-specific foot orthoses (Experimental): Morpho-specific thermo-molded foot orthoses are designed according to the patient's morphotype.
  Orthoses are custom-molded from different materials such as BIOFLUX resin, Covercuir MF, EVA300/60, EVA400/70, PE255/55, ABSORB Dur and CAPITON PU.
  Interventions: Device: Foot orthoses
- Placebo foot orthoses (Placebo Comparator): The placebo foot orthoses will be made with the same principle of molding and with the same materials as for the experimental group. The only difference is that they involve no active corrective insert element : they will be made without morphotype correction.
  Interventions: Device: Foot orthoses

INTERVENTIONS:
Device: Foot orthoses

SUMMARY:
Patellofemoral pain syndrome is one of the most common musculoskeletal disorders. It is defined as an anterior knee pain. Its origin is a conflict during patellar tracking, due to patellofemoral malalignment and soft tissue overload.

A few recent studies seem to show a benefit of prefabricated feet orthoses in patellofemoral pain syndrome, alone or in association with rehabilitation. However, no one has analyzed the outcome of morpho-specific foot orthoses in a prospective randomized study.

The purpose of this prospective randomized study is to compare clinical outcomes in daily living and in sports activities, between morpho-specific and placebo foot orthoses.

Morpho-specific foot orthoses are designed according to the patient's morphotype. They are intended to correct structural defects of the hindfoot, midfoot and forefoot, in the aim to correct abnormal overload during patellofemoral tracking.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 12-40 years
* Patellofemoral pain syndrome
* Patient affiliated to a social protection regime
* Patient who signed an informed consent
* For teenagers with no complete growth and muscular maturation, failure of appropriate rehabilitation during minimum 2 months
* Patient informed of the results of the prior medical examination
* Normality (no sign of osteoarthritis) of the knee radiographs
* Ability to read and understand French

Exclusion Criteria:

* Knee osteoarthritis
* Systemic disease
* Inflammatory rheumatism disease
* Unstable knee
* Prior patellofemoral dislocation
* Osteochondrosis
* Referred pain from a hip or spine disease (particularly proximal femoral epiphysiolysis in the teenagers)
* A history of patellar trauma
* A history of knee surgery
* Meniscus, ligament or osteochondral pathology
* Knee tendinitis or bursitis
* Neurologic disease
* Pregnancy
* Antidepressant therapy or behavioral disorder
* Patient unable to comply the required maximum observance
* Impossibility to give enlightened information to the patient
* Patient under guardianship

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Item Pain of the KOOS Score | Twice : at inclusion and at 10 weeks follow-up with feet orthoses

SECONDARY OUTCOMES:
KOOS Score (items Symptoms, Activities of daily living, Sport and recreation function, Knee-related quality of life) | Twice : at inclusion and at 10 weeks follow-up with feet orthoses
Kujala Score | Twice : at inclusion and at 10 weeks follow-up with feet orthoses
Pain level | Twice : at inclusion and at 10 weeks follow-up with feet orthoses
  Visual Analog Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Cabinet libéral - 12, rue du Puits, Haguenau
  - Service de Chirurgie Orthopédique - Hôpital CCOM - Hôpitaux Universitaires de Strasbourg, Illkirch-Graffenstaden
  - Cabinet libéral - 50, avenue des Vosges, Strasbourg